CLINICAL TRIAL: NCT07132619
Title: Effect of Hypothermic Total Circulatory Arrest Duration on Renal Function in Pulmonary Endarterectomy Surgery: A Retrospective Single-Center Study
Brief Title: Kidney Injury After PTE: Association With Hypothermic Circulatory Arrest Duration
Status: Completed | Type: Observational
Sponsor: Ebru Girgin Dinc (Other)
Responsible Party: Sponsor-Investigator, Ebru Girgin Dinc, M.D., Anesthesiologist, Koşuyolu Kartal Heart Training and Research Hospital
Organization: Koşuyolu Kartal Heart Training and Research Hospital (Other)
Other Study IDs: HTCA-PEA
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Acute Kidney Failure; Pulmonary Thromboembolisms; Hypothermic Circulatory Arrest Time
Keywords: AKI; Acute Kıdney Injury; PTE; Pulmonary Thromboembolisms; TCA; Hypothermic Circulatory Arrest Time
MeSH Terms: conditions — Acute Kidney Injury; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective, single-center observational study evaluates the association between the duration of total circulatory arrest (TCA) and the incidence and severity of postoperative acute kidney injury (AKI) in patients undergoing pulmonary endarterectomy between 2018 and 2020. AKI will be classified according to KDIGO 2012 criteria, using both changes in serum creatinine and hourly urine output tracked over 48 hours. The study aims to determine the frequency of AKI, its association with TCA duration, and to identify potential perioperative risk factors contributing to renal dysfunction. Secondary outcomes will include the relationship between AKI and in-hospital mortality, length of intensive care unit stay, and total hospital length of stay. Findings from this study may provide insights into optimizing intraoperative management strategies to reduce postoperative renal morbidity in patients undergoing pulmonary endarterectomy.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common and clinically significant complication following cardiothoracic surgery, particularly in procedures requiring circulatory arrest. Pulmonary endarterectomy (PEA), which is often performed under deep hypothermic total circulatory arrest (TCA), carries a notable risk for postoperative renal dysfunction due to ischemia-reperfusion injury and intraoperative hemodynamic instability. The reported incidence of AKI after PEA varies widely, ranging from 20% to 50%, and is associated with increased morbidity, prolonged hospitalization, and elevated mortality. Despite this clinical importance, few studies have systematically evaluated AKI in the setting of PEA using both serum creatinine and urine output criteria.

The 2012 Kidney Disease: Improving Global Outcomes (KDIGO) guidelines emphasize the use of both biomarkers in AKI diagnosis, yet most studies rely solely on creatinine. Given the limitations of isolated creatinine-based assessment, integrating hourly urine output offers a more comprehensive understanding of renal function. This study was designed to evaluate the relationship between TCA duration and the incidence and severity of AKI in patients undergoing PEA, using full KDIGO 2012 criteria. The goal was to better characterize AKI risk in this high-acuity population and inform perioperative management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-85 years
* Underwent pulmonary endarterectomy between 2018 and 2020

Exclusion Criteria:

* Age below 18 years
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients aged 18 to 85 years who underwent pulmonary endarterectomy at the Cardiothoracic Surgery Unit of Kosuyolu Kartal Heart Training and Research Hospital (Kosuyolu KHTRH), a single tertiary referral center in Istanbul, Turkey, between January 1, 2018, and December 31, 2020. Patients meeting the inclusion criteria will have complete perioperative data available, including total circulatory arrest duration and postoperative renal function parameters. Individuals younger than 18 years of age and pregnant women at the time of surgery will be excluded.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Association Between Total Circulatory Arrest Duration and Incidence of Postoperative Acute Kidney Injury | up to 48 hours, postoperatively
  The presence or absence of postoperative acute kidney injury (AKI) will be determined according to KDIGO 2012 criteria, based on both changes in serum creatinine and hourly urine output within the first 48 hours after surgery. The primary measure will be the relationship between total circulatory arrest (TCA) duration (in minutes) and the occurrence of AKI, analyzed as a binary variable (yes/no).

SECONDARY OUTCOMES:
Severity of Acute Kidney Injury According to KDIGO Staging | up to 48 hours, postoperatively
  Severity of postoperative acute kidney injury (AKI) will be graded according to KDIGO 2012 criteria (Stages 1-3) using both changes in serum creatinine and hourly urine output within the first 48 hours after surgery.
Length of Intensive Care Unit Stay | up to 30 days postoperatively
  Total number of days from the date of ICU admission immediately following surgery until discharge from the ICU.
In-Hospital Mortality | up to 30 days postoperatively
  Death from any cause during the same hospitalization as the index pulmonary endarterectomy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Atakan ERKILINC, MD, Associate Professor, Principal Investigator — University of Health Sciences, Kosuyolu Heart Training and Research Hospital, Kartal, ISTANBUL
Locations (1):
- Kosuyolu Heart Training and Research Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol